CLINICAL TRIAL: NCT00046839
Title: A Phase I/II Trial of a COX-2 Inhibitor, Celebrex (Celecoxib), [National Screening Committee# 719627] With Limited Field Radiation for Intermediate Prognosis Patients With Locally Advanced Non-Small Cell Lung Cancer, With Analysis of Prognostic Factors
Brief Title: Celecoxib and Radiation Therapy in Treating Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0213; CDR0000069476
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Cyclooxygenase 2 Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I: Celecoxib 200mg BID + RT (Experimental): COX-2 Inhibitor: Celecoxib 200 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
  Interventions: Drug: celecoxib; Radiation: radiation therapy
- Phase I: Celecoxib 400mg BID + RT (Experimental): COX-2 Inhibitor: Celecoxib 400 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
  Interventions: Drug: celecoxib; Radiation: radiation therapy
- Phase II: Celecoxib 400mg BID + RT (Experimental): COX-2 Inhibitor: Celecoxib 400 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
  Interventions: Drug: celecoxib; Radiation: radiation therapy

INTERVENTIONS:
Drug: celecoxib
  Other Names: COX-2 Inhibitor
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Celecoxib may stop the growth of tumor cells by stopping blood flow to the tumor and may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I/II trial to study the effectiveness of combining celecoxib with radiation therapy in treating patients who have locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and the recommended phase II dose of concurrent celecoxib and limited-field radiotherapy in intermediate-prognosis patients with locally advanced non-small cell lung cancer.
* Determine the efficacy and toxicity of this regimen in these patients.
* Determine how the predictors of mortality in the general population (i.e., comorbid conditions, functional status, quality of life, and psychological status) influence prognosis, toxicity, and outcomes of therapy in patients treated with this regimen.
* Correlate circulating levels of vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), and interleukin-8 (IL8) with survival in patients treated with this regimen.
* Correlate circulating levels of interleukin-1 (IL1), interleukin-6 (IL6), and transforming growth factor-beta (TGFB) with pulmonary toxicity in patients treated with this regimen.

OUTLINE: This is a phase I dose-escalation study of celecoxib followed by a phase II, multicenter study.

* Phase I: Patients receive oral celecoxib twice daily. Beginning on day 6, patients undergo thoracic radiotherapy 5 days a week for 3-6.5 weeks . Patients continue to receive celecoxib for up to 2 years in the absence of disease progression or unacceptable toxicity.
* Phase II: If fewer than 3 of the first 6 patients experience dose-limiting toxicity, then the dose of celecoxib is escalated for all patients in the study, including those in the first cohort.

Quality of life is assessed at baseline and at 3, 6, and 12 months after start of therapy.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-12 patients will be accrued for the phase I portion of this study and a total of 116 patients will be accrued for the phase II portion of this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Inoperable stage IIB OR
  * Unresectable stage IIIA or IIIB
  * No evidence of hematogenous metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 2 AND more than 5% weight loss over the past 3 months OR
* Zubrod 0-1 AND less than 5% weight loss over the past 3 months and refuses chemotherapy or are medically unable to tolerate combined modality therapy

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2 times upper limit of normal
* International Normalized Ratio (INR) no greater than 3.0 if taking warfarin

Renal

* Creatinine clearance at least 50 mL/min

Other

* No active gastrointestinal ulcers or bleeding within the past 3 months
* No other malignancy within the past 3 years except nonmelanoma skin cancer
* No known hypersensitivity to celecoxib
* No prior allergic-type reactions to sulfonamides
* No prior asthma, urticaria, or allergic-type reactions to aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior neoadjuvant chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* No prior thoracic radiotherapy

Surgery

* No prior complete or subtotal tumor resection

Other

* No concurrent NSAIDs, lithium, furosemide, or angiotensin-converting enzyme inhibitors
* Concurrent aspirin (325 mg/day) for cardioprotection allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-07; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Gore, MD, Study Chair — Medical College of Wisconsin
Locations (44):
- United States (44):
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Mount Holly, New Jersey
  - Albuquerque Regional Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - North Star Lodge Cancer Center, Yakima, Washington
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - University of Wisconsin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin

REFERENCES:
- [Result] Gore E, Bae K, Langer C, Extermann M, Movsas B, Okunieff P, Videtic G, Choy H. Phase I/II trial of a COX-2 inhibitor with limited field radiation for intermediate prognosis patients who have locally advanced non-small-cell lung cancer: radiation therapy oncology group 0213. Clin Lung Cancer. 2011 Mar;12(2):125-30. doi: 10.1016/j.cllc.2011.03.007. Epub 2011 Apr 11. PMID 21550559

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Phase I: Celecoxib 200mg BID + RT: COX-2 Inhibitor: Celecoxib 200 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
- Experimental: Phase I/II: Celecoxib 400mg BID + RT: COX-2 Inhibitor: Celecoxib 400 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
Period: Overall Study
Arm/Group | Experimental: Phase I: Celecoxib 200mg BID + RT | Experimental: Phase I/II: Celecoxib 400mg BID + RT
Started | 8 | 13
Completed | 7 (Subjects contributing data to either primary analysis are considered to have completed the study.) | 11 (Subjects contributing data to either primary analysis are considered to have completed the study.)
Not Completed | 1 | 2
Not completed — Ineligible / No protocol treatment | 0 | 2
Not completed — Withdrawal of consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Phase I: Celecoxib 200mg BID + RT | Experimental: Phase I/II: Celecoxib 400mg BID + RT | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 88] | 71 [47 to 82] | 72 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Celecoxib Combined With Radiation Therapy (RT)
Description: Patients were followed for at least 90 days from start of RT and carefully evaluated with respect to treatment morbidity. A dose limiting toxicity (DLT) was defined as grade 3 or 4 nonhematologic (excluding nausea, vomiting, and alopecia) and grade 4 hematologic toxicities. Six patients were to be accrued at each dose level. If no more than three of the six patients experienced a DLT then that dose level was considered acceptable and dose escalation occurred by accruing six more patients at the next dose level. Otherwise, the preceding dose level, if any, would be declared the MTD. The MTD would be used for the Phase II arm. At a given dose, the probability of halting dose escalation when the true toxicity is 50% or higher is at least 66% (power). In addition, if the true DLT rate is instead 20%, there will still be a 10% probability of halting dose escalation at a given dose level (type I error).
  Rating scale: 0 = not the MTD, 1 = MTD
Time Frame: Start of treatment to 90 days
Population: The first six eligible patients who started protocol treatment at each dose level.
Measure: Number; unit: units on a scale
Groups:
- Phase I: Celecoxib 200mg BID + RT: COX-2 Inhibitor: Celecoxib 200 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
  celecoxib
  radiation therapy
- Phase I: Celecoxib 400mg BID + RT: COX-2 Inhibitor: Celecoxib 400 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
  celecoxib
  radiation therapy
Arm/Group | Phase I: Celecoxib 200mg BID + RT | Phase I: Celecoxib 400mg BID + RT
Number analyzed (Participants) | 6 | 6
units on a scale | 0 | 1

2. Primary Outcome: Overall Survival
Description: Because only 21 patients (18 analyzable) out of 128 planned were accrued on this study, all analyzable patients were combined to report overall survival. The original study design planned for a comparison to a historical control, but due to the small number of patients, survival time is only reported, not tested.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 12 months.
Population: Eligible patients who started protocol treatment.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Experimental: Phase I/II: Celecoxib 200 or 400mg BID + RT: COX-2 Inhibitor: Celecoxib 200 or 400 mg b.i.d, 7 days/week begins 5 days prior to start of radiation therapy (RT). Once RT begins, Celecoxib a.m. dose 1-2 hours prior to RT. Administer for 2 years or until disease progression.
  Concurrent Radiation Therapy: 2 Gy daily, 30-33 fractions, 5 days/week for 6-7 weeks, for a total dose of 60-66 Gy; or 3 Gy daily, 15 fractions, 5 days/week for 3-4 weeks for a total dose of 45 Gy.
Arm/Group | Experimental: Phase I/II: Celecoxib 200 or 400mg BID + RT
Number analyzed (Participants) | 18
years | 10.0 [6.1 to 16.7]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given SAE (serious adverse event) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Arm/Group | Experimental: Phase I: Celecoxib 200mg BID + RT | Experimental: Phase I/II: Celecoxib 400mg BID + RT
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/11
Other Adverse Events (participants affected / at risk) | 7/7 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Phase I: Celecoxib 200mg BID + RT (N=7) | Experimental: Phase I/II: Celecoxib 400mg BID + RT (N=11)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 | 0
Infection without neutropenia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Phase I: Celecoxib 200mg BID + RT (N=7) | Experimental: Phase I/II: Celecoxib 400mg BID + RT (N=11)
Hematologic-Other (Blood and lymphatic system disorders) | 2 | 0
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2 | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 | 0
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 3 | 0
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 1 | 1
Dysphagia-pharyngeal related to radiation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Edema (General disorders) | 0 | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 4 | 4
Late RT Toxicity: Lung (General disorders) | 2 | 1
Late RT Toxicity: Other (General disorders) | 1 | 0
Late RT Toxicity: Skin (within the irradiated field) (General disorders) | 1 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 3 | 3
Creatinine (Investigations) | 3 | 0
Leukocytes (total WBC) (Investigations) | 1 | 0
Lymphopenia (Investigations) | 1 | 0
Metabolic-Other (Investigations) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 0
SGPT (ALT) (Investigations) | 2 | 0
Weight loss (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Neuropathy motor (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Renal/GU-Other (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This study stopped accrual early with 21 subjects accrued out of 128 planned, therefore only the phase I and phase II primary outcomes were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No